CLINICAL TRIAL: NCT04146883
Title: Post-procedure Antibiotic Prophylaxis for Cardiac Electrical Device Implantation: ABxFREE Study
Acronym: ABxFREE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Ju-Yi Chen, Associate Professor, Department of Internal Medicine, College of Medicine, National Cheng Kung University, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B-ER-108-130
Record Dates: First submitted 2019-10-25; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Post Procedural Infection; Pacemaker Electrode Infection; Antibiotics; Implantable Defibrillator User
Keywords: Prophylactic antibiotics; Cardiac implantable electronic device infection
MeSH Terms: interventions — Anti-Bacterial Agents; Cephalexin

STUDY DESIGN:
Intervention Model Description: This study is a multi-center, prospective, randomized and open-labeled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post procedural antibiotics treatment (Experimental): This group was treated with pre-procedural (pacemaker or ICD implantation) prophylactic once intravenous antibiotics (cefazolin 1000mg or else if allergy to cefazolin) and post procedural oral prophylactic antibiotics
  Interventions: Drug: Antibiotics
- Pre procedural antibiotics treatment only (No Intervention): This group was only treated with pre-procedural (pacemaker or ICD implantation) prophylactic once intravenous antibiotics (cefazolin 1000mg or else if allergy to cefazolin).

INTERVENTIONS:
Drug: Antibiotics — Post-procedural one-day iv cefazolin then 3-day prophylactic cephalexin
  Other Names: Cephalexin
  Arms: Post procedural antibiotics treatment

SUMMARY:
This study is a multi-center open-label randomized study, and we sought to investigate the redundancy of post-procedural prophylactic antibiotics in cardiac implantable electronic device implantation. There are 2 arms in this study. One arm will receive pre-procedural intravenous antibiotics only. The other arm will receive both pre-procedural intravenous antibiotics and post-procedural 3-day oral antibiotics.

DETAILED DESCRIPTION:
There is general agreement on the benefits of preoperative prophylactic antibiotics which had been documented in previous studies. Concerns of bacterial resistance and unnecessary cost, our prospective observational case-control study had suggested the redundancy of post-procedural antibiotics. In this well-designed study, we sought to investigate the efficacy of post-procedural antibiotics and confirm the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for permanent pacemaker or implantable cardioverter defibrillator implantation according to current guidelines

Exclusion Criteria:

* Hospitalization for more than 7 days
* End stage renal disease with hemodialysis or peritonealysis
* Patients receive cardiac resynchronization therapy, His-bundle pacemaker, leadless pacemaker, or sub-cutaneous implantable cardioverter defibrillator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-08-19 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac implantable electronic device related infection | 1 year
  Any local and systemic signs/symptoms (pocket erosion, localized pocket erythema, swelling, heatness, pain, fever, bacteremia, lead/valvular vegetation) will be monitored during follow-up. The definition and classification of CIED related infection are based on the current guideline and expert consensus statement.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Yi Chen, PhD, Principal Investigator — National Cheng-Kung Univerity Hospital
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
We will not share IPD due to the restriction of NCKUH IRB.

REFERENCES:
- [Background] Sandoe JA, Barlow G, Chambers JB, Gammage M, Guleri A, Howard P, Olson E, Perry JD, Prendergast BD, Spry MJ, Steeds RP, Tayebjee MH, Watkin R; British Society for Antimicrobial Chemotherapy; British Heart Rhythm Society; British Cardiovascular Society; British Heart Valve Society; British Society for Echocardiography. Guidelines for the diagnosis, prevention and management of implantable cardiac electronic device infection. Report of a joint Working Party project on behalf of the British Society for Antimicrobial Chemotherapy (BSAC, host organization), British Heart Rhythm Society (BHRS), British Cardiovascular Society (BCS), British Heart Valve Society (BHVS) and British Society for Echocardiography (BSE). J Antimicrob Chemother. 2015 Feb;70(2):325-59. doi: 10.1093/jac/dku383. Epub 2014 Oct 29. PMID 25355810
- [Background] Kusumoto FM, Schoenfeld MH, Wilkoff BL, Berul CI, Birgersdotter-Green UM, Carrillo R, Cha YM, Clancy J, Deharo JC, Ellenbogen KA, Exner D, Hussein AA, Kennergren C, Krahn A, Lee R, Love CJ, Madden RA, Mazzetti HA, Moore JC, Parsonnet J, Patton KK, Rozner MA, Selzman KA, Shoda M, Srivathsan K, Strathmore NF, Swerdlow CD, Tompkins C, Wazni O. 2017 HRS expert consensus statement on cardiovascular implantable electronic device lead management and extraction. Heart Rhythm. 2017 Dec;14(12):e503-e551. doi: 10.1016/j.hrthm.2017.09.001. Epub 2017 Sep 15. No abstract available. PMID 28919379
- [Result] Lee WH, Huang TC, Lin LJ, Lee PT, Lin CC, Lee CH, Chao TH, Li YH, Chen JY. Efficacy of postoperative prophylactic antibiotics in reducing permanent pacemaker infections. Clin Cardiol. 2017 Aug;40(8):559-565. doi: 10.1002/clc.22698. Epub 2017 Apr 26. PMID 28444977
- [Result] Chiang KH, Chao TF, Lee WS, Lin YJ, Tuan TC, Kong CW. How Long Should Prophylactic Antibiotics be Prescribed for Permanent Pacemaker Implantations? One Day versus Three Days. Acta Cardiol Sin. 2013 Jul;29(4):341-6. PMID 27122728
- [Result] Madadi S, Kafi M, Kheirkhah J, Azhari A, Kiarsi M, Mehryar A, Fazelifar A, Alizadehdiz A, Emkanjoo Z, Haghjoo M. Postoperative antibiotic prophylaxis in the prevention of cardiac implantable electronic device infection. Pacing Clin Electrophysiol. 2019 Feb;42(2):161-165. doi: 10.1111/pace.13592. Epub 2019 Jan 4. PMID 30575054
- [Result] de Oliveira JC, Martinelli M, Nishioka SA, Varejao T, Uipe D, Pedrosa AA, Costa R, D'Avila A, Danik SB. Efficacy of antibiotic prophylaxis before the implantation of pacemakers and cardioverter-defibrillators: results of a large, prospective, randomized, double-blinded, placebo-controlled trial. Circ Arrhythm Electrophysiol. 2009 Feb;2(1):29-34. doi: 10.1161/CIRCEP.108.795906. Epub 2009 Feb 10. PMID 19808441